CLINICAL TRIAL: NCT05868382
Title: A Phase 2, Randomized, Active-Controlled, Observer-Blind, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA Vaccine Candidate Variations in Healthy Adults 18 to 49 Years of Age
Brief Title: Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA Vaccine Candidate Variations in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-CRID-004
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Influenza
Keywords: mRNA-1010; Influenza Vaccine; Moderna
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1010 influenza vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- mRNA-1010 Dose C (Experimental): Participants will receive a single dose of mRNA-1010 by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1010
- mRNA-1010.4 Dose B (Experimental): Participants will receive a single dose of mRNA-1010.4 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010.4
- mRNA-1010.4 Dose C (Experimental): Participants will receive a single dose of mRNA-1010.4 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010.4
- mRNA-1010.6 Dose A (Experimental): Participants will receive a single dose of mRNA-1010.6 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010.6
- mRNA-1010.6 Dose B (Experimental): Participants will receive a single dose of mRNA-1010.6 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010.6
- mRNA-1010.6 Dose C (Experimental): Participants will receive a single dose of mRNA-1010.6 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010.6

INTERVENTIONS:
Biological: mRNA-1010 — Sterile liquid for injection
  Arms: mRNA-1010 Dose C
Biological: mRNA-1010.4 — Sterile liquid for injection
  Arms: mRNA-1010.4 Dose B; mRNA-1010.4 Dose C
Biological: mRNA-1010.6 — Sterile liquid for injection
  Arms: mRNA-1010.6 Dose A; mRNA-1010.6 Dose B; mRNA-1010.6 Dose C

SUMMARY:
The main purpose of the study is to evaluate the safety, reactogenicity, and the immunogenicity of mRNA-1010 vaccine candidate variations.

ELIGIBILITY:
Inclusion Criteria:

* Investigator has assessed that the participant understands and is willing and physically able to comply with protocol mandated follow up, including all procedures.
* For assigned females at birth and of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, and agreement to continue adequate contraception through 90 days following vaccine administration.

Exclusion Criteria:

* Participant has had close contact with someone with laboratory-confirmed influenza infection or with someone who has been treated with antiviral therapies for influenza (for example, Tamiflu®) within the past 5 days prior to Day 1.
* Participant is acutely ill or febrile (temperature ≥38.0℃elcius [100.4°Fahrenheit]) 72 hours prior to or at the Screening visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day screening window.
* Participant has a history of a diagnosis or condition that, in the judgment of the investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Reported history of congenital or acquired immunodeficiency, immunosuppressive condition or immune-mediated disease, asplenia, or recurrent severe infections.
* Participant has tested positive for influenza by local health authority-approved testing methods within 150 days prior to Day 1.
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of mRNA vaccines or any components of the mRNA-1010 or influenza vaccines, including egg protein.
* Participant has received systemic immunosuppressants for >14 days in total within 180 days prior to Day 1 (for corticosteroids, ≥10 mg/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study. Inhaled, nasal and topical steroids are allowed. Intra-articular and epidural steroid injections are not allowed within 28 days before and/or after study intervention dosing.
* Participant has received any vaccine authorized or approved by local health agency ≤28 days prior to study intervention dosing (Day 1) or plans to receive a vaccine authorized or approved by local health agency within 28 days before or after study intervention dosing.
* Participant has received a licensed seasonal influenza vaccine within 5 months (150 days) prior to Day 1.
* Participant has participated in any investigational seasonal influenza vaccine study within12 months prior to Day 1.
* Participant is not aware whether they have received an influenza vaccine in the prior 12 months.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to Day 1 or plans to donate blood products during the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - CenExel RCA, Hollywood, Florida
  - Suncoast Research Group, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Rockville Internal Medicine, Rockville, Maryland
  - DM Clinical Research, Southfield, Michigan
  - Meridian Clinical Research, Hastings, Nebraska
  - Meridian Clinical Research, Lincoln, Nebraska
  - United Medical Associates, Binghamton, New York
  - DM Clinical Research, Sugar Land, Texas
  - Texas Center for Drug Development, Tomball, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- mRNA-1010: Participants received a single dose of mRNA-1010 by intramuscular (IM) injection on Day 1.
- mRNA-1010.4 Low Dose: Participants received mRNA-1010.4 at a low dose level by IM injection on Day 1.
- mRNA-1010.4 High Dose: Participants received mRNA-1010.4 at a high dose level by IM injection on Day 1.
- mRNA-1010.6 Low Dose: Participants received mRNA-1010.6 at a low dose level by IM injection on Day 1.
- mRNA-1010.6 Medium Dose: Participants received mRNA-1010.6 at a medium dose level by IM injection on Day 1.
- mRNA-1010.6 High Dose: Participants received mRNA-1010.6 at a high dose level by IM injection on Day 1.
Period: Overall Study
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
Started | 60 | 30 | 60 | 30 | 30 | 60
Received Injection | 60 | 30 | 60 | 30 | 30 | 60
Safety Set (All participants who received 1 dose of study intervention. Participants were included in the study arm corresponding to the study intervention that they received.) | 60 | 30 | 60 | 30 | 31 (1 participant randomized to receive mRNA-1010.6 High Dose but actually received mRNA-1010.6 Medium Dose.) | 59 (1 participant randomized to receive mRNA-1010.6 High Dose but actually received mRNA-1010.6 Medium Dose.)
Solicited Safety Set (All participants who received 1 dose of study intervention and contributed any solicited AR data (that is, had at least 1 post baseline solicited safety [eDiary] assessment). Participants were included in the study arm corresponding to the study intervention that they received.) | 60 | 30 | 60 | 30 | 31 (1 participant randomized to receive mRNA-1010.6 High Dose but actually received mRNA-1010.6 Medium Dose.) | 59 (1 participant randomized to receive mRNA-1010.6 High Dose but actually received mRNA-1010.6 Medium Dose.)
Per-Protocol Set (All randomized participants who received the study intervention, complied with the injection schedule, timing of immunogenicity blood sampling to have a baseline (Day 1), had at least 1 post injection assessment, had a Day 29 assessment that was within 22 days to 43 days after injection, had no important protocol deviations which impacted the immune response, and did not use prohibited medication or nonstudy vaccines against influenza.) | 55 | 28 | 56 | 29 | 28 | 52
Completed | 54 | 30 | 54 | 26 | 27 | 54
Not Completed | 6 | 0 | 6 | 4 | 3 | 6
Not completed — Lost to Follow-up | 5 | 0 | 6 | 4 | 2 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants who received the study intervention.
Groups:
- mRNA-1010: Participants received a single dose of mRNA-1010 by IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose | Total
Number analyzed (Participants) | 60 | 30 | 60 | 30 | 30 | 60 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.08) | 36.7 (8.06) | 34.6 (7.87) | 36.7 (9.05) | 35.9 (7.56) | 33.8 (7.54) | 35.0 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 17 | 40 | 13 | 17 | 31 | 152
  Male | 26 | 13 | 20 | 17 | 13 | 29 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 6 | 25 | 7 | 12 | 19 | 87
  Not Hispanic or Latino | 39 | 24 | 33 | 21 | 18 | 40 | 175
  Unknown or Not Reported | 3 | 0 | 2 | 2 | 0 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Asian | 2 | 2 | 4 | 0 | 0 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 24 | 12 | 17 | 14 | 10 | 17 | 94
  White | 29 | 14 | 35 | 14 | 18 | 37 | 147
  More than one race | 4 | 1 | 1 | 0 | 1 | 1 | 8
  Unknown or Not Reported | 1 | 1 | 3 | 1 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were collected in an electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. All solicited ARs considered causally related to injection were graded 0-4 (per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials); lower score indicates lower severity, and a higher score indicates greater severity. Note, not all solicited ARs were considered adverse events (AEs). The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set included all participants who received 1 dose of study intervention and contributed any solicited AR data (that is, had at least 1 post baseline solicited safety [eDiary] assessment). Participants were included in the study intervention group corresponding to the study intervention that they received.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
Number analyzed (Participants) | 60 | 30 | 60 | 30 | 31 | 59
Participants
  Any | 50 | 27 | 53 | 18 | 25 | 55
  Grade 1 | 22 | 11 | 11 | 11 | 12 | 15
  Grade 2 | 24 | 11 | 32 | 5 | 12 | 34
  Grade 3 | 4 | 5 | 10 | 2 | 1 | 6
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was an AE that was not solicited using a participant diary and that was communicated by a participant who has signed the informed consent. An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. Number of participants with unsolicited AEs (SAEs and non-serious AEs) up to 28 days post-vaccination are reported in this outcome measure.
Time Frame: Up to 28 days post-vaccination
Population: Safety Set included all participants who received 1 dose of study intervention. Participants were included in the study arm corresponding to the study intervention that they received.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
Number analyzed (Participants) | 60 | 30 | 60 | 30 | 31 | 59
Participants | 11 | 4 | 9 | 0 | 4 | 7

3. Primary Outcome: Number of Participants With SAEs, AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Study or Treatment Discontinuation
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that lead to an unscheduled visit to an healthcare practitioner. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or coronavirus disease 2019 [COVID-19] and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). Number of participants with SAEs, AESIs, MAAEs, and AEs leading to discontinuation up to the end of study (Day 181) are reported in this outcome measure.
Time Frame: Day 1 to Day 181 (end of study [EOS])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
Number analyzed (Participants) | 60 | 30 | 60 | 30 | 31 | 59
Participants
  SAEs | 1 | 0 | 2 | 1 | 0 | 1
  AESIs | 0 | 0 | 0 | 0 | 0 | 0
  MAAEs | 14 | 5 | 12 | 2 | 3 | 8
  AEs Leading to Study or Treatment Discontinuation | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies, as Measured by Hemagglutination Inhibition (HAI) Assay for Vaccine-matched Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. 95% CI was calculated based on the t-distribution of log-transformed values for GM titer, then back transformed to original scale for presentation.
Time Frame: Days 1 (Baseline), 8, 29, 91, and 181
Population: Per-Protocol Set: all randomized participants who received study drug, complied with injection schedule, timing of immunogenicity blood sampling to have a baseline (Day 1), had at least 1 post injection assessment, had a Day 29 assessment that was within 22 days to 43 days after injection, had no important protocol deviations which impacted immune response, and did not use prohibited medication/nonstudy vaccines against influenza. 'Number analyzed'= participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
Number analyzed (Participants) | 55 | 28 | 56 | 29 | 28 | 52
titer
  Influenza A H1N1 Antibody: Day 1 | 52.4 [41.5 to 66.2] | 60.9 [41.9 to 88.7] | 72.9 [53.9 to 98.5] | 78.2 [54.5 to 112.1] | 50.5 [34.2 to 74.6] | 48.2 [36.7 to 63.3]
  Influenza A H1N1 Antibody: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza A H1N1 Antibody: Day 8 | 226.2 [164.8 to 310.6] | 272.4 [196.2 to 378.3] | 337.2 [244.9 to 464.3] | 240.2 [163.8 to 352.2] | 259.3 [166.9 to 403.0] | 331.3 [247.0 to 444.5]
  Influenza A H1N1 Antibody: Day 29 | 334.4 [247.8 to 451.2] | 316.1 [214.5 to 465.8] | 394.9 [299.1 to 521.5] | 255.0 [177.7 to 366.1] | 269.1 [184.5 to 392.5] | 349.0 [266.9 to 456.3]
  Influenza A H1N1 Antibody: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza A H1N1 Antibody: Day 91 | 168.9 [125.2 to 227.8] | 202.4 [144.2 to 284.2] | 229.3 [174.4 to 301.4] | 160.0 [108.8 to 235.4] | 174.5 [117.0 to 260.3] | 179.6 [137.8 to 234.1]
  Influenza A H1N1 Antibody: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza A H1N1 Antibody: Day 181 | 127.6 [95.9 to 169.7] | 164.1 [119.9 to 224.7] | 167.8 [122.4 to 230.0] | 119.9 [82.4 to 174.5] | 123.8 [88.2 to 173.8] | 137.4 [106.1 to 177.9]
  Influenza A H3N2 Antibody: Day 1 | 33.3 [26.3 to 42.3] | 46.4 [31.6 to 68.1] | 41.2 [32.8 to 51.9] | 37.2 [26.7 to 51.9] | 29.7 [21.5 to 40.9] | 27.4 [21.8 to 34.4]
  Influenza A H3N2 Antibody: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza A H3N2 Antibody: Day 8 | 125.6 [88.7 to 178.1] | 187.9 [128.2 to 275.5] | 188.4 [147.5 to 240.6] | 109.1 [71.4 to 166.6] | 125.0 [80.0 to 195.2] | 162.3 [118.2 to 222.8]
  Influenza A H3N2 Antibody: Day 29 | 159.0 [115.8 to 218.4] | 262.7 [170.9 to 403.8] | 248.2 [192.2 to 320.6] | 124.4 [78.2 to 198.1] | 136.2 [89.7 to 206.9] | 160.0 [118.7 to 215.7]
  Influenza A H3N2 Antibody: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza A H3N2 Antibody: Day 91 | 105.1 [77.3 to 142.7] | 146.8 [101.4 to 212.6] | 154.8 [116.6 to 205.5] | 99.5 [69.8 to 141.9] | 94.0 [66.9 to 132.0] | 103.6 [80.0 to 134.0]
  Influenza A H3N2 Antibody: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza A H3N2 Antibody: Day 181 | 87.8 [66.0 to 116.8] | 124.9 [84.6 to 184.2] | 107.9 [81.7 to 142.3] | 68.2 [46.4 to 100.4] | 67.7 [48.3 to 94.8] | 87.0 [65.2 to 116.2]
  Influenza B/ Victoria Lineage: Day 1 | 63.4 [55.1 to 72.9] | 78.1 [60.5 to 100.9] | 82.5 [66.9 to 101.8] | 74.5 [59.4 to 93.4] | 64.0 [49.8 to 82.3] | 67.8 [58.2 to 78.9]
  Influenza B/ Victoria Lineage: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza B/ Victoria Lineage: Day 8 | 88.9 [72.2 to 109.3] | 164.0 [119.5 to 225.1] | 194.7 [145.8 to 260.0] | 150.7 [112.2 to 202.4] | 129.6 [91.9 to 182.8] | 126.4 [100.7 to 158.7]
  Influenza B/ Victoria Lineage: Day 29 | 94.3 [75.4 to 117.8] | 174.5 [124.2 to 245.3] | 218.0 [160.3 to 296.5] | 132.2 [99.2 to 176.2] | 120.4 [90.3 to 160.6] | 132.8 [104.2 to 169.3]
  Influenza B/ Victoria Lineage: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza B/ Victoria Lineage: Day 91 | 89.2 [77.2 to 103.2] | 126.5 [100.9 to 158.5] | 138.2 [109.6 to 174.2] | 100.9 [78.2 to 130.1] | 84.1 [66.4 to 106.5] | 94.2 [80.8 to 109.7]
  Influenza B/ Victoria Lineage: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza B/ Victoria Lineage: Day 181 | 62.9 [53.7 to 73.7] | 75.2 [56.2 to 100.5] | 83.9 [68.5 to 102.7] | 59.9 [47.2 to 76.1] | 60.3 [49.7 to 73.2] | 60.2 [51.8 to 69.9]
  Influenza B/ Yamagata Lineage: Day 1 | 71.9 [57.6 to 89.7] | 107.7 [72.3 to 160.4] | 96.3 [75.6 to 122.8] | 99.2 [70.0 to 140.5] | 77.1 [57.3 to 103.6] | 84.9 [67.4 to 106.9]
  Influenza B/ Yamagata Lineage: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza B/ Yamagata Lineage: Day 8 | 181.2 [142.0 to 231.1] | 293.5 [195.8 to 440.0] | 305.7 [233.2 to 400.8] | 198.3 [141.9 to 277.3] | 215.5 [155.2 to 299.2] | 367.6 [280.4 to 481.8]
  Influenza B/ Yamagata Lineage: Day 29 | 181.5 [146.6 to 224.7] | 275.8 [187.5 to 405.8] | 336.2 [270.4 to 418.1] | 205.7 [142.4 to 297.0] | 187.9 [136.8 to 258.2] | 309.5 [246.8 to 388.1]
  Influenza B/ Yamagata Lineage: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza B/ Yamagata Lineage: Day 91 | 134.1 [112.7 to 159.5] | 190.3 [140.0 to 258.7] | 218.9 [173.4 to 276.2] | 160.0 [120.1 to 213.2] | 141.4 [107.8 to 185.5] | 194.8 [161.7 to 234.7]
  Influenza B/ Yamagata Lineage: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza B/ Yamagata Lineage: Day 181 | 109.4 [91.3 to 131.2] | 137.9 [101.0 to 188.3] | 140.6 [113.6 to 174.1] | 111.6 [79.5 to 156.4] | 125.4 [98.6 to 159.4] | 138.3 [114.3 to 167.4]

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-HA Antibodies, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% confidence interval (CI) for GMFR was calculated based on the t distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Baseline, Days 8, 29, 91, and 181
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
Number analyzed (Participants) | 55 | 28 | 56 | 29 | 28 | 52
ratio
  Influenza A H1N1 Antibody: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza A H1N1 Antibody: Day 8 | 4.27 [3.13 to 5.783] | 4.47 [2.95 to 6.78] | 4.38 [3.18 to 6.04] | 3.07 [2.04 to 4.64] | 5.13 [3.40 to 7.75] | 6.87 [4.79 to 9.86]
  Influenza A H1N1 Antibody: Day 29 | 6.38 [4.58 to 8.89] | 5.19 [3.37 to 7.99] | 5.42 [3.94 to 7.44] | 3.26 [2.15 to 4.95] | 5.32 [3.31 to 8.57] | 7.24 [5.16 to 10.17]
  Influenza A H1N1 Antibody: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza A H1N1 Antibody: Day 91 | 3.13 [2.36 to 4.17] | 3.32 [2.34 to 4.71] | 3.08 [2.24 to 4.25] | 2.05 [1.50 to 2.81] | 3.45 [1.94 to 6.13] | 3.71 [2.69 to 5.13]
  Influenza A H1N1 Antibody: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza A H1N1 Antibody: Day 181 | 2.36 [1.80 to 3.10] | 2.69 [1.88 to 3.86] | 2.23 [1.61 to 3.08] | 1.59 [1.14 to 2.21] | 2.43 [1.43 to 4.12] | 2.87 [2.12 to 3.88]
  Influenza A H3N2 Antibody: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza A H3N2 Antibody: Day 8 | 3.82 [2.87 to 5.08] | 4.05 [3.03 to 5.42] | 4.44 [3.46 to 5.71] | 2.93 [2.05 to 4.19] | 4.21 [2.82 to 6.29] | 6.11 [4.65 to 8.02]
  Influenza A H3N2 Antibody: Day 29 | 4.77 [3.74 to 6.09] | 5.66 [3.98 to 8.06] | 6.02 [4.68 to 7.75] | 3.34 [2.27 to 4.91] | 4.59 [3.08 to 6.83] | 5.85 [4.49 to 7.61]
  Influenza A H3N2 Antibody: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza A H3N2 Antibody: Day 91 | 3.11 [2.47 to 3.93] | 3.17 [2.20 to 4.55] | 3.79 [2.81 to 5.12] | 2.76 [1.91 to 3.99] | 3.17 [2.14 to 4.69] | 3.76 [3.05 to 4.65]
  Influenza A H3N2 Antibody: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza A H3N2 Antibody: Day 181 | 2.59 [2.06 to 3.26] | 2.69 [2.01 to 3.61] | 2.66 [1.99 to 3.55] | 2.06 [1.43 to 2.97] | 2.25 [1.60 to 3.16] | 3.14 [2.47 to 4.00]
  Influenza B/Victoria Lineage: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza B/Victoria Lineage: Day 8 | 1.41 [1.20 to 1.65] | 2.10 [1.53 to 2.88] | 2.39 [1.93 to 3.00] | 2.02 [1.59 to 2.58] | 2.03 [1.62 to 2.52] | 1.90 [1.58 to 2.30]
  Influenza B/Victoria Lineage: Day 29 | 1.49 [1.26 to 1.76] | 2.23 [1.65 to 3.03] | 2.64 [2.11 to 3.31] | 1.78 [1.40 to 2.26] | 1.88 [1.54 to 2.29] | 1.96 [1.61 to 2.38]
  Influenza B/Victoria Lineage: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza B/Victoria Lineage: Day 91 | 1.36 [1.16 to 1.59] | 1.62 [1.27 to 2.06] | 1.65 [1.38 to 1.97] | 1.34 [1.04 to 1.73] | 1.31 [1.04 to 1.66] | 1.39 [1.19 to 1.64]
  Influenza B/Victoria Lineage: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza B/Victoria Lineage: Day 181 | 0.95 [0.79 to 1.15] | 0.96 [0.75 to 1.24] | 0.98 [0.81 to 1.19] | 0.74 [0.55 to 0.99] | 0.93 [0.74 to 1.15] | 0.89 [0.73 to 1.09]
  Influenza B/Yamagata Lineage: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza B/Yamagata Lineage: Day 8 | 2.53 [2.02 to 3.17] | 2.73 [2.04 to 3.65] | 3.20 [2.42 to 4.23] | 2.00 [1.49 to 2.68] | 2.80 [2.07 to 3.78] | 4.32 [3.41 to 5.47]
  Influenza B/Yamagata Lineage: Day 29 | 2.53 [2.04 to 3.12] | 2.56 [1.99 to 3.29] | 3.49 [2.72 to 4.48] | 2.07 [1.75 to 2.74] | 2.44 [1.75 to 3.39] | 3.65 [2.90 to 4.59]
  Influenza B/Yamagata Lineage: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza B/Yamagata Lineage: Day 91 | 1.83 [1.54 to 2.17] | 1.77 [1.42 to 2.20] | 2.21 [1.78 to 2.74] | 1.59 [1.24 to 2.03] | 1.83 [1.37 to 2.46] | 2.29 [1.88 to 2.80]
  Influenza B/Yamagata Lineage: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza B/Yamagata Lineage: Day 181 | 1.47 [1.24 to 1.75] | 1.28 [0.97 to 1.69] | 1.41 [1.13 to 1.76] | 1.09 [0.84 to 1.42] | 1.61 [1.22 to 2.13] | 1.63 [1.34 to 1.97]

6. Secondary Outcome: Percentage of Participants With Seroresponse for mRNA-1010, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Seroresponse was defined as (a) a post-vaccination antibody titer ≥ 4 * lower limit of quantification (LLOQ) if baseline (Day 1) antibody titer was < LLOQ or (b) a post-vaccination antibody titer ≥ 4-fold of baseline antibody titer if baseline antibody titer was ≥ LLOQ.
Time Frame: Days 8, 29, 91, and 181
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
Number analyzed (Participants) | 55 | 28 | 56 | 29 | 28 | 52
percentage of participants
  Influenza A H1N1 Antibody: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza A H1N1 Antibody: Day 8 | 54.7 [40.4 to 68.4] | 50.0 [30.6 to 69.4] | 50.9 [36.8 to 64.9] | 31.0 [15.3 to 50.8] | 60.7 [40.6 to 78.5] | 70.0 [55.4 to 82.1]
  Influenza A H1N1 Antibody: Day 29 | 69.1 [55.2 to 80.9] | 53.6 [33.9 to 72.5] | 60.7 [46.8 to 73.5] | 41.4 [23.5 to 61.1] | 60.7 [40.6 to 78.5] | 69.2 [54.9 to 81.3]
  Influenza A H1N1 Antibody: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza A H1N1 Antibody: Day 91 | 58.8 [44.2 to 72.4] | 50.0 [30.6 to 69.4] | 38.5 [25.3 to 53.0] | 29.6 [13.8 to 50.2] | 42.9 [24.5 to 62.8] | 51.0 [36.6 to 65.2]
  Influenza A H1N1 Antibody: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza A H1N1 Antibody: Day 181 | 36.5 [23.6 to 51.0] | 39.3 [21.5 to 59.4] | 31.4 [19.1 to 45.9] | 16.7 [4.7 to 37.4] | 37.0 [19.4 to 57.6] | 42.0 [28.2 to 56.8]
  Influenza A H3N2 Antibody: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza A H3N2 Antibody: Day 8 | 54.7 [40.4 to 68.4] | 67.9 [47.6 to 84.1] | 56.6 [42.3 to 70.2] | 41.4 [23.5 to 61.1] | 57.1 [37.2 to 75.5] | 70.0 [55.4 to 82.1]
  Influenza A H3N2 Antibody: Day 29 | 65.5 [51.4 to 77.8] | 67.9 [47.6 to 84.1] | 73.2 [59.7 to 84.2] | 58.6 [38.9 to 76.5] | 64.3 [44.1 to 81.4] | 69.2 [54.9 to 81.3]
  Influenza A H3N2 Antibody: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza A H3N2 Antibody: Day 91 | 54.9 [40.3 to 68.9] | 50.0 [30.6 to 69.4] | 57.7 [43.2 to 71.3] | 40.7 [22.4 to 61.2] | 60.7 [40.6 to 78.5] | 56.9 [42.2 to 70.7]
  Influenza A H3N2 Antibody: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza A H3N2 Antibody: Day 181 | 42.3 [28.7 to 56.8] | 35.7 [18.6 to 55.9] | 45.1 [31.1 to 59.7] | 25.0 [9.8 to 46.7] | 37.0 [19.4 to 57.6] | 48.0 [33.7 to 62.6]
  Influenza B/Victoria Lineage: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza B/Victoria Lineage: Day 8 | 11.3 [4.3 to 23.0] | 17.9 [6.1 to 36.9] | 28.3 [16.8 to 42.3] | 20.7 [8.0 to 39.7] | 17.9 [6.1 to 36.9] | 18.0 [8.6 to 31.4]
  Influenza B/Victoria Lineage: Day 29 | 12.7 [5.3 to 24.5] | 25.0 [10.7 to 44.9] | 35.7 [23.4 to 49.6] | 17.2 [5.8 to 35.8] | 14.3 [4.0 to 32.7] | 19.2 [9.6 to 32.5]
  Influenza B/Victoria Lineage: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza B/Victoria Lineage: Day 91 | 3.9 [0.5 to 13.5] | 14.3 [4.0 to 32.7] | 17.3 [8.2 to 30.3] | 11.1 [2.4 to 29.2] | 3.6 [0.1 to 18.3] | 3.9 [0.5 to 13.5]
  Influenza B/Victoria Lineage: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza B/Victoria Lineage: Day 181 | 5.8 [1.2 to 15.9] | 7.1 [0.9 to 23.5] | 3.9 [0.5 to 13.5] | 4.2 [0.1 to 21.1] | 0 [0.0 to 12.8] | 4.0 [0.5 to 13.7]
  Influenza B/Yamagata Lineage: Day 8: number analyzed (Participants) | 53 | 28 | 53 | 29 | 28 | 50
  Influenza B/Yamagata Lineage: Day 8 | 35.8 [23.1 to 50.2] | 39.3 [21.5 to 59.4] | 39.6 [26.5 to 54.0] | 20.7 [8.0 to 39.7] | 28.6 [13.2 to 48.7] | 62.0 [47.2 to 75.3]
  Influenza B/Yamagata Lineage: Day 29 | 29.1 [17.6 to 42.9] | 32.1 [15.9 to 52.4] | 50.0 [36.3 to 63.7] | 27.6 [12.7 to 47.2] | 25.0 [10.7 to 44.9] | 53.8 [39.5 to 67.8]
  Influenza B/Yamagata Lineage: Day 91: number analyzed (Participants) | 51 | 28 | 52 | 27 | 28 | 51
  Influenza B/Yamagata Lineage: Day 91 | 17.6 [8.4 to 30.9] | 14.3 [4.0 to 32.7] | 26.9 [15.6 to 41.0] | 14.8 [4.2 to 33.7] | 21.4 [8.3 to 41.0] | 31.4 [19.1 to 45.9]
  Influenza B/Yamagata Lineage: Day 181: number analyzed (Participants) | 52 | 28 | 51 | 24 | 27 | 50
  Influenza B/Yamagata Lineage: Day 181 | 11.5 [4.4 to 23.4] | 10.7 [2.3 to 28.2] | 11.8 [4.4 to 23.9] | 4.2 [0.1 to 21.1] | 11.1 [2.4 to 29.2] | 16.0 [7.2 to 29.1]

ADVERSE EVENTS:
Time Frame: Day 1 up to the end of study (Day 181)
Description: All-cause mortality and AE (Serious and Non-serious) data were collected and reported for all randomized participants.
  Participants were included in the study arm corresponding to the study intervention that they received.
Arm/Group | mRNA-1010 | mRNA-1010.4 Low Dose | mRNA-1010.4 High Dose | mRNA-1010.6 Low Dose | mRNA-1010.6 Medium Dose | mRNA-1010.6 High Dose
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/30 | 0/60 | 0/30 | 0/31 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/30 | 2/60 | 1/30 | 0/31 | 1/59
Other Adverse Events (participants affected / at risk) | 0/60 | 0/30 | 0/60 | 0/30 | 0/31 | 3/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mRNA-1010 (N=60) | mRNA-1010.4 Low Dose (N=30) | mRNA-1010.4 High Dose (N=60) | mRNA-1010.6 Low Dose (N=30) | mRNA-1010.6 Medium Dose (N=31) | mRNA-1010.6 High Dose (N=59)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mRNA-1010 (N=60) | mRNA-1010.4 Low Dose (N=30) | mRNA-1010.4 High Dose (N=60) | mRNA-1010.6 Low Dose (N=30) | mRNA-1010.6 Medium Dose (N=31) | mRNA-1010.6 High Dose (N=59)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT05868382/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT05868382/SAP_001.pdf